CLINICAL TRIAL: NCT02142140
Title: Efficacy of Careful Medication and Tailored Case Management Follow up Treatment for Children With Attention Deficit Hyperactivity Disorder
Brief Title: Follow up Treatment of Children With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Lily Hechtman, Professor of Psychiatry and Pediatrics; Director of Research - Division of Child Psychiatry, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOP 123412
Record Dates: First submitted 2014-05-14; First posted 2014-05-20 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: Treatment of ADHD; Long-term treatment follow-up
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride; Methylphenidate; Lisdexamfetamine Dimesylate; Adderall; Dextroamphetamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medication Monitoring & Case Management (Experimental): All children entered into this study will be prescribed medication for their ADHD symptoms (usually a long-acting stimulant). Based on the individual needs of the child and family, they could receive the following interventions - Academic and organization skills, social skills training and parent training. Participants randomized to this group will meet with the study clinicians 4 times a year for medication monitoring and adjustment. This group will also receive a monthly call from a case manager who will explore the child's academic, social and emotional functioning. Depending on the needs of the child and family, the case manager may offer 1 to 5 intervention sessions with the child (e.g. social skills, anger management), the family (e.g. family counselling), and the school (e.g. consultation with the teacher).
  Interventions: Behavioral: Academic and Organization skills; Behavioral: Parent Training; Behavioral: Social Skills Training; Drug: Long-acting stimulant
- Community Follow-up Group (Active Comparator): All children entered into this study will be prescribed medication for their ADHD symptoms (usually a long-acting stimulant). Based on the individual needs of the child and family, they could receive the following interventions - Academic and organization skills, social skills training and parent training. Families randomized to this group will be referred to their pediatricians or family physicians for medication follow-up and their local Community Health Clinic (CLSC) for other psychosocial interventions that may be required and available.
  Interventions: Behavioral: Academic and Organization skills; Behavioral: Parent Training; Behavioral: Social Skills Training; Drug: Long-acting stimulant

INTERVENTIONS:
Behavioral: Academic and Organization skills — This program aims at teaching children organization, time management and stress management skills. They are also taught academic strategies in reading, writing, and math. The program consists of six, 90 minute sessions.
Behavioral: Parent Training — The Parent Training Program: The parent training program is designed to increase parental understanding of ADHD; establish attentive, positive interactions, and solve problems collaboratively. Eight weekly group sessions lasting about 2 hours each will be conducted by trained psychologists, social workers, or clinical nurses. Homework assignments and detailed summary sheets will be used to promote technique acquisition and generalization.
Behavioral: Social Skills Training — Social Skills and Anger Management Training: The social skills training program is based on understanding yourself and others, and being able to understand things from the other's perspective. The program uses direct instruction, modelling, behavioural rehearsal, feedback, and social reinforcement. The following are covered: joining in, understanding emotions, dealing with anger, using self-control, responding to teasing / bullying, and staying out of fights.
Drug: Long-acting stimulant — The medication prescribed is usually a long-acting stimulant that is carefully titrated to the child's optimal dose (normally that dose above which further improvement is not seen and side effects are manageable). Once optimal dose is reached, children are followed at regular once per three month visits for medication monitoring. In this group the child can be referred for a medication reevaluation and adjustment as many times as is needed.
  Other Names: Biphentin; Strattera; Concerta; Ritalin; Vyvanse; Adderall; Dexedrine
  Arms: Medication Monitoring & Case Management
Drug: Long-acting stimulant — The medication prescribed is usually a long-acting stimulant that is carefully titrated to the child's optimal dose (normally that dose above which further improvement is not seen and side effects are manageable). Once optimal dose is reached, children are followed by their pediatrician, with a frequency at his/her discretion.
  Other Names: Biphentin; Strattera; Concerta; Ritalin; Vyvanse; Adderall; Dexedrine
  Arms: Community Follow-up Group

SUMMARY:
The purpose of the study is to examine how well two types of treatment follow up work compared to one another:

1. standard community follow up
2. medication monitoring plus tailored case management follow up.

A child's participation will involve 3 months of treatment consisting of medication and psychological, behavioural, and academic interventions tailored to their individual needs.

Following this treatment, the child will be randomly assigned to receive two years of either community follow up or medication monitoring plus tailored case management follow up delivered by the study team. During both types of follow up, at 6 month intervals, the parent and child will be asked to complete interviews with our study personnel and comprehensive assessments pertaining to ADHD symptoms and various other areas of functioning.

Parents will also be asked to obtain information from the child's teacher regarding the child's functioning at 6 month intervals during the school year.

ELIGIBILITY:
Inclusion Criteria:

* age 6 to 12 years
* DSM-IV ADHD diagnosis by a specialist i.e. child psychiatrist or developmental paediatrician (DSM 5 ADHD criteria do not differ dramatically from DSM IV criteria for children)
* Intelligence Quotient (IQ) > 80 as per the Wechsler Intelligence Scale for Children (WISC-IV)
* Proficiency in English or French

Exclusion Criteria:

* History of Autism Spectrum Disorder (ASD) or psychosis
* Significant brain traumas (encephalitis, head injury requiring hospitalization, etc.)
* Major medical conditions or impairments that would interfere with the ability of the child to complete testing or take psychostimulants, e.g., epilepsy, cardiac abnormalities, or renal abnormalities.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 326 (Estimated)
Dates: Start 2012-12; Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Attention Deficit Hyperactivity Disorder (ADHD) symptomatology (measured via Conners' Global Index - Parent and Teacher Version) | At baseline - no medication
Attention Deficit Hyperactivity Disorder (ADHD) symptomatology (measured via Conners' Global Index - Parent and Teacher Version) | Following 3 months of tailored treatment (including medication)
Attention Deficit Hyperactivity Disorder (ADHD) symptomatology (measured via Conners' Global Index - Parent and Teacher Version) | Six months after tailored treatment ends - on medication
Attention Deficit Hyperactivity Disorder (ADHD) symptomatology (measured via Conners' Global Index - Parent and Teacher Version) | Twelve months after tailored treatment has ended - on medication
Attention Deficit Hyperactivity Disorder (ADHD) symptomatology (measured via Conners' Global Index - Parent and Teacher Version) | Eighteen months after tailored treatment has ended - on medication
Attention Deficit Hyperactivity Disorder (ADHD) symptomatology (measured via Conners' Global Index - Parent and Teacher Version) | Twenty-four months after tailored treatment has ended - on medication

SECONDARY OUTCOMES:
Social skills (measured via Parent and Teacher Social Skills Rating Scale) | At baseline - no medication
Academic achievement (measured via Wechsler Individual Achievement Test (WIAT)) | At baseline - no medication
Emotional and symptomatic functioning (measured via the Achenbach Child Behavior Check List (CBCL)) | At baseline - no medication
Overall functioning (measured via the Weiss Functional Impairment Scale (WFIRS)) | At baseline - no medication
Overall functioning (measured via the Clinical Global Impression Scale (CGI)) | Assessed at baseline
Social skills (measured via Parent and Teacher Social Skills Rating Scale) | Following 3 months of tailored treatment (including medication)
Social skills (measured via Parent and Teacher Social Skills Rating Scale) | Six months after tailored treatment ends - on medication
Social skills (measured via Parent and Teacher Social Skills Rating Scale) | Twelve months after tailored treatment has ended - on medication
Social skills (measured via Parent and Teacher Social Skills Rating Scale) | Eighteen months after tailored treatment has ended - on medication
Social skills (measured via Parent and Teacher Social Skills Rating Scale) | Twenty-four months after tailored treatment has ended - on medication
Academic achievement (measured via Wechsler Individual Achievement Test (WIAT)) | Twelve month after tailored treatment has ended - on medication
Academic achievement (measured via Wechsler Individual Achievement Test (WIAT)) | Twenty-four months after tailored treatment has ended
Emotional and symptomatic functioning (measured via the Achenbach Child Behavior Check List (CBCL)) | Following 3 months of tailored treatment (including medication)
Emotional and symptomatic functioning (measured via the Achenbach Child Behavior Check List (CBCL)) | Six months after tailored treatment ends - on medication
Emotional and symptomatic functioning (measured via the Achenbach Child Behavior Check List (CBCL)) | Twelve months after tailored treatment has ended - on medication
Emotional and symptomatic functioning (measured via the Achenbach Child Behavior Check List (CBCL)) | Eighteen months after tailored treatment has ended - on medication
Emotional and symptomatic functioning (measured via the Achenbach Child Behavior Check List (CBCL)) | Twenty-four months after tailored treatment has ended - on medication
Overall functioning (measured via the Weiss Functional Impairment Scale (WFIRS)) | Following 3 months of tailored treatment (including medication)
Overall functioning (measured via the Weiss Functional Impairment Scale (WFIRS)) | Six months after tailored treatment ends - on medication
Overall functioning (measured via the Weiss Functional Impairment Scale (WFIRS)) | Twelve months after tailored treatment has ended - on medication
Overall functioning (measured via the Weiss Functional Impairment Scale (WFIRS)) | Eighteen months after tailored treatment has ended - on medication
Overall functioning (measured via the Weiss Functional Impairment Scale (WFIRS)) | Twenty-four months after tailored treatment has ended - on medication
Overall functioning (measured via the Clinical Global Impression Scale (CGI)) | Following 3 months of tailored treatment (including medication)
Overall functioning (measured via the Clinical Global Impression Scale (CGI)) | Three months after tailored treatment ends - on medication
  For participants randomized to the medication monitoring and tailored case management follow-up group.
Overall functioning (measured via the Clinical Global Impression Scale (CGI)) | Six months after tailored treatment ends - on medication
  For participants randomized to the medication monitoring and tailored case management follow-up group.
Overall functioning (measured via the Clinical Global Impression Scale (CGI)) | Nine months after tailored treatment ends - on medication
  For participants randomized to the medication monitoring and tailored case management follow-up group.
Overall functioning (measured via the Clinical Global Impression Scale (CGI)) | Twelve months after tailored treatment ends - on medication
  For participants randomized to the medication monitoring and tailored case management follow-up group.
Overall functioning (measured via the Clinical Global Impression Scale (CGI)) | Fifteen months after tailored treatment ends - on medication
  For participants randomized to the medication monitoring and tailored case management follow-up group.
Overall functioning (measured via the Clinical Global Impression Scale (CGI)) | Eighteen months after tailored treatment ends - on medication
  For participants randomized to the medication monitoring and tailored case management follow-up group.
Overall functioning (measured via the Clinical Global Impression Scale (CGI)) | Twenty-one months after tailored treatment ends - on medication
  For participants randomized to the medication monitoring and tailored case management follow-up group.
Overall functioning (measured via the Clinical Global Impression Scale (CGI)) | Twenty-four months after tailored treatment ends - on medication
  For participants randomized to the medication monitoring and tailored case management follow-up group.

CONTACTS AND LOCATIONS:
Overall Officials: Lily Hechtman, MD, FRCPC, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Natalie Grizenko, MD, FRCPC, Principal Investigator — Douglas Mental Health University Institute; Ridha Joober, MD, PhD, Principal Investigator — Douglas Mental Health University Institute
Locations (2):
- Canada (2):
  - Montreal Children's Hospital, Montreal, Quebec
  - Douglas Mental Health University Institute, Montreal, Quebec